CLINICAL TRIAL: NCT01155115
Title: Inflammatory and Microbiologic Markers in Sputum in Response to Pulmonary Exacerbation: Comparing Cystic Fibrosis With Primary Ciliary Dyskinesia
Brief Title: Inflammatory and Microbiologic Markers in Sputum: Comparing Cystic Fibrosis With Primary Ciliary Dyskinesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Felix Ratjen, Division Head, Respiratory Medicine, The Hospital for Sick Children
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000013966
Record Dates: First submitted 2010-06-29; First posted 2010-07-01 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Cystic Fibrosis; Primary Ciliary Dyskinesia
Keywords: pediatrics; CF; PCD; exacerbation; inflammatory markers; induced sputum
MeSH Terms: conditions — Cystic Fibrosis; Ciliary Motility Disorders | interventions — Respiratory Physiological Phenomena

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Primary Ciliary Dyskinesia (PCD) Patients (Experimental)
  Interventions: Procedure: Sputum Collection; Procedure: Pulmonary Function Testing; Procedure: Exhaled Nitric Oxide
- Cystic Fibrosis (CF) Patients (Experimental)
  Interventions: Procedure: Sputum Collection; Procedure: Pulmonary Function Testing; Procedure: Exhaled Nitric Oxide

INTERVENTIONS:
Procedure: Sputum Collection — Each study participant will be invited to expectorate sputum for culture, sensitivity, cytology and analysis of cytokine levels. Culture and sensitivity will be performed routinely at the beginning of a pulmonary exacerbation, as per standard of care, and will only be performed at subsequent visits if there is clinical indication. A volume of 5ml of sputum will be required at each visit for analysis. If the participant is unable to expectorate this volume of sputum, he/she will be invited to induce sputum instead as per standard protocols.
Procedure: Pulmonary Function Testing — Participants will perform spirometry at each visit according to the American Thoracic Society and European Respiratory Society guidelines.
Procedure: Exhaled Nitric Oxide — The investigators will measure exhaled Nitric Oxide (eNO) at each visit according to the American Thoracic Society and European Respiratory Society guidelines using a chemiluminescence analyzer. Briefly, single breath exhalation are performed in triplicate at flows of 30, 50, 100, 150, 200 and 250 ml/s and eNO is measured at the end of the exhalation. The higher the flow rate the more peripheral the airways that are being sampled.

SUMMARY:
The objective of this study is to compare the lower airways inflammatory response to infection/pulmonary exacerbation among children known to have Primary Ciliary Dyskinesia (PCD) with children known to have Cystic Fibrosis (CF) as measured by the presence of inflammatory mediators in expectorated/induced sputum.

DETAILED DESCRIPTION:
The inflammatory response to infection and pulmonary exacerbation in CF is well documented, as is the response to intravenous antibiotic treatment. On the other hand, the inflammatory response to infection and treatment in PCD has not been well characterized. Given differences in disease progression, we hypothesize that children with CF respond to infection with a more exaggerated and prolonged inflammatory response than those with PCD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Cystic Fibrosis (CF) as defined by two or more clinical features of CF and a documented sweat chloride > 60 mEq/L by quantitative pilocarpine iontophoresis test or a genotype showing two well characterized disease-causing mutations or a diagnosis of Primary Ciliary Dyskinesia (PCD) as follows: definite PCD (compatible phenotype, diagnostic abnormality of ciliary ultrastructure and/or two disease-causing gene mutations) or "probable" PCD (compatible phenotype, ciliary biopsy not diagnostic but low nasal NO (<100nl/min) with negative investigation screen for both CF and immunodeficiency
* Informed consent and verbal assent (as appropriate) provided by the subject's parent or legal guardian and the subject
* 6-18 years of age at enrolment and able to perform reproducible spirometry
* Clinically stable at enrolment (FEV > 30%, oxyhaemoglobin sats > 93%)
* Ability to comply with study visits and study procedures

Exclusion Criteria:

* Respiratory culture positive for non-tuberculous mycobacteria (NTM), Stenotrophomonas maltophilia, Aspergillus fumigatus, Burkholderia cepacia complex, or Pseudomonas aeruginosa within past year.
* Use of intravenous antibiotics or oral quinolones within previous 14 days
* Use of inhaled antibiotics within the previous 28 days
* Pneumothorax or haemoptysis

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2010-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Change in sputum bacterial colony count | Up to 100 days
  For the following organisms (Staphylococcus aureus, Haemophilus influenza) in response to a prescribed treatment course of oral antibiotics.
  Colony count will be done at three time points:
  * during respiratory exacerbation (Visit 1 - Day 0),
  * post-antibiotic treatment of exacerbation (Visit 2 - Day 21-42),
  * and on return to clinical baseline (Visit 3 - Day 42-100 (End of Study)).during the study.
Airway Inflammatory Profile | Up to 100 days
  As measured by sputum interleukin 8 (IL-8) at three time points:
  * during respiratory exacerbation (Visit 1 - Day 0),
  * post-antibiotic treatment of exacerbation (Visit 2 - Day 21-42),
  * and on return to clinical baseline (Visit 3 - Day 42-100 (End of Study)).

SECONDARY OUTCOMES:
Culture, identification, and antibiotic susceptibility pattern of respiratory pathogens from sputum samples | Up to 100 days
  Will be done at three time points:
  * during respiratory exacerbation (Visit 1 - Day 0),
  * post-antibiotic treatment of exacerbation (Visit 2 - Day 21-42),
  * and on return to clinical baseline (Visit 3 - Day 42-100 (End of Study)).during the study.
Tolerability and need for sputum induction in Cystic Fibrosis (CF) patients in comparison to Primary Ciliary Dyskinesia (PCD) patients | Up to 100 days
  Sputum will be collected at three time points:
  * during respiratory exacerbation (Visit 1 - Day 0),
  * post-antibiotic treatment of exacerbation (Visit 2 - Day 21-42),
  * and on return to clinical baseline (Visit 3 - Day 42-100 (End of Study)).
Change in forced expiratory volume in 1 second (FEV1) in response to a treatment course of antibiotics for pulmonary exacerbation. | Up to 100 days
  FEV1 will be measured at three time points:
  * during respiratory exacerbation (Visit 1 - Day 0),
  * post-antibiotic treatment of exacerbation (Visit 2 - Day 21-42),
  * and on return to clinical baseline (Visit 3 - Day 42-100 (End of Study)).during the study.
Other markers of airway inflammation | Up to 100 days
  Measurement of sputum white cell and neutrophil count (absolute and relative values), neutrophil elastase, nitric oxide (NO), NO metabolites and arginase levels at three time points:
  * during respiratory exacerbation (Visit 1 - Day 0),
  * post-antibiotic treatment of exacerbation (Visit 2 - Day 21-42),
  * and on return to clinical baseline (Visit 3 - Day 42-100 (End of Study)).

CONTACTS AND LOCATIONS:
Overall Officials: Felix Ratjen, MD, Principal Investigator — The Hospital for Sick Children, Toronto Canada
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Grasemann H, McDonald N, Yuan XZ, Dell S, Waters V, Ratjen F. Lower Airway Nitrogen Oxide Levels in Children with Primary Ciliary Dyskinesia Is Linked to Neutrophilic Inflammation. J Pediatr. 2022 May;244:230-233. doi: 10.1016/j.jpeds.2022.01.040. Epub 2022 Feb 2. PMID 35120987
- [Derived] Ratjen F, Waters V, Klingel M, McDonald N, Dell S, Leahy TR, Yau Y, Grasemann H. Changes in airway inflammation during pulmonary exacerbations in patients with cystic fibrosis and primary ciliary dyskinesia. Eur Respir J. 2016 Mar;47(3):829-36. doi: 10.1183/13993003.01390-2015. Epub 2015 Nov 19. PMID 26585432